CLINICAL TRIAL: NCT01659619
Title: Effect of Erythromycin Before Endoscopy of Patients With Subtotal Gastrectomy (STG), High Risk of Gastric Stasis : Randomized and Prospective Study
Brief Title: Effect of Erythromycin Before Endoscopy of Patients With Subtotal Gastrectomy (STG), High Risk of Gastric Stasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Myung-gui Choi, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KC12MISI0164
Record Dates: First submitted 2012-04-10; First posted 2012-08-08 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Subtotal Gastrectomy; Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Erythromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- erythromycin (Experimental)
  Interventions: Drug: Erythromycin
- saline (No Intervention)

INTERVENTIONS:
Drug: Erythromycin — 125mg in normal saline single use infusion for 5 min.
  Arms: erythromycin

SUMMARY:
Erythromycin has a prokinetic effect through Motilin receptor. It evokes migrating motor complex with longer and stronger contraction.

In patients with upper gastrointestinal bleeding, It has been shown that erythromycin could clear the stomach of blood, so visual examination could be improved.

Frequent food stasis is encounted when we examine patients with subtotal gastrectomy. It is postulated that erythromycin reduce food stasis and help to improve endoscopy in these cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergone STG (billroth I, billroth II, R-Y STG) within 5 years to treat gastric cancer
* Stage of T1-2N0M0

Exclusion Criteria:

* concomitant therapy with astemizole, cisapride, dihydroergotamine, ergotamine, pimozide, or terfenadine, narcotics, alpha-2-adrenergic agonist, TCA, CCB, dopamine agonist, muscarinic cholinergic antagonists, octreotide, exenatide and GLP-1 agonist, phenothiazines
* chemotherapy Hx.
* hypersensitivity to erythromycin or any component of the product
* pregnancy or lactation
* comobidity : DM, AIDS, neurologic disease(parkinsonism, multiple sclerosis, brainstem stroke or tumor, diabetic or amyloid neuropathy, or primary dysautonomias) scleroderma and other connective tissue disease, recent viral enteritis history
* recurrence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
degree of food stasis | when endoscopy is performed.
  ref> Gastric Cancer (2002) 5: 83-89

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Gyu Choi, M.D., Principal Investigator — Department of Internal Medicine, College of Medicine, The Catholic University of Korea, Seoul, Republic of Korea
Locations (1):
- Seoul St. Mary hospital, Seoul, South Korea

REFERENCES:
- [Background] Sarna SK, Soergel KH, Koch TR, Stone JE, Wood CM, Ryan RP, Arndorfer RC, Cavanaugh JH, Nellans HN, Lee MB. Gastrointestinal motor effects of erythromycin in humans. Gastroenterology. 1991 Dec;101(6):1488-96. doi: 10.1016/0016-5085(91)90383-v. PMID 1955115
- [Background] Annese V, Janssens J, Vantrappen G, Tack J, Peeters TL, Willemse P, Van Cutsem E. Erythromycin accelerates gastric emptying by inducing antral contractions and improved gastroduodenal coordination. Gastroenterology. 1992 Mar;102(3):823-8. doi: 10.1016/0016-5085(92)90164-t. PMID 1537520
- [Background] Bruley des Varannes S, Parys V, Ropert A, Chayvialle JA, Roze C, Galmiche JP. Erythromycin enhances fasting and postprandial proximal gastric tone in humans. Gastroenterology. 1995 Jul;109(1):32-9. doi: 10.1016/0016-5085(95)90266-x. PMID 7797033
- [Background] Ramirez B, Eaker EY, Drane WE, Hocking MP, Sninsky CA. Erythromycin enhances gastric emptying in patients with gastroparesis after vagotomy and antrectomy. Dig Dis Sci. 1994 Nov;39(11):2295-300. doi: 10.1007/BF02087641. PMID 7956594
- [Background] Kendall BJ, Chakravarti A, Kendall E, Soykan I, McCallum RW. The effect of intravenous erythromycin on solid meal gastric emptying in patients with chronic symptomatic post-vagotomy-antrectomy gastroparesis. Aliment Pharmacol Ther. 1997 Apr;11(2):381-5. doi: 10.1046/j.1365-2036.1997.148324000.x. PMID 9146779
- [Background] Frossard JL, Spahr L, Queneau PE, Giostra E, Burckhardt B, Ory G, De Saussure P, Armenian B, De Peyer R, Hadengue A. Erythromycin intravenous bolus infusion in acute upper gastrointestinal bleeding: a randomized, controlled, double-blind trial. Gastroenterology. 2002 Jul;123(1):17-23. doi: 10.1053/gast.2002.34230. PMID 12105828
- [Background] Altraif I, Handoo FA, Aljumah A, Alalwan A, Dafalla M, Saeed AM, Alkhormi A, Albekairy AK, Tamim H. Effect of erythromycin before endoscopy in patients presenting with variceal bleeding: a prospective, randomized, double-blind, placebo-controlled trial. Gastrointest Endosc. 2011 Feb;73(2):245-50. doi: 10.1016/j.gie.2010.09.043. Epub 2010 Dec 8. PMID 21145052
- [Background] Kubo M, Sasako M, Gotoda T, Ono H, Fujishiro M, Saito D, Sano T, Katai H. Endoscopic evaluation of the remnant stomach after gastrectomy: proposal for a new classification. Gastric Cancer. 2002;5(2):83-9. doi: 10.1007/s101200200014. PMID 12111583
- [Derived] Jun BY, Choi MG, Lee JY, Baeg MK, Moon SJ, Lim CH, Kim JS, Cho YK, Lee IS, Kim SW, Choi KY. Premedication with erythromycin improves endoscopic visualization of the gastric mucosa in patients with subtotal gastrectomy: a prospective, randomized, controlled trial. Surg Endosc. 2014 May;28(5):1641-7. doi: 10.1007/s00464-013-3364-y. Epub 2014 Jan 1. PMID 24380989